CLINICAL TRIAL: NCT05308134
Title: MaxiMoM: Individualized Fortification of Human Milk for Infants Born ≤ 1250 g; a Three Arm Randomized Clinical Trial
Brief Title: Individualized Fortification of Human Milk for Infants Born ≤ 1250 g (MaxiMoM-InForM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1861
Record Dates: First submitted 2021-11-10; First posted 2022-04-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Very Low Birth Weight Infant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard fortification (Active Comparator)
  Interventions: Other: Standard fortification
- Target fortification (Experimental)
  Interventions: Other: Target fortification
- BUN adjustable fortification (Experimental)
  Interventions: Other: BUN adjustable fortification

INTERVENTIONS:
Other: Standard fortification — Standard fortification assumes that the nutrient content of human milk is constant and involves use of a standard fixed dose of multi-nutrient fortifier and as appropriate nutrient modulars.
  Arms: Standard fortification
Other: Target fortification — Target fortification involves use of a multi-nutrient fortifier as well as weekly analysis of energy and macronutrients of human milk and subsequent addition of fat and protein modulars if needed.
  Arms: Target fortification
Other: BUN adjustable fortification — BUN (blood urea nitrogen) adjustable fortification involves use of a multi-nutrient fortifier as well as weekly BUN tests and subsequent addition of a protein modular according to a prescribed algorithm.
  Arms: BUN adjustable fortification

SUMMARY:
Very low birth weight infants have increased nutritional needs. Extra nutrients are added to their human milk feeds to help improve their nutritional status, growth and neurodevelopment. Standard fortification of human milk is routine in most neonatal units in North America, but despite the added nutrients, infants are often discharged from hospitals with poor growth, and their neurodevelopment remains suboptimal. Two individualized fortification methods, target and BUN adjustable, have been proposed to improve the nutrient supply to infants. However, there is currently insufficient evidence to support the implementation of individualized fortification or one method over the other. Therefore, this study will randomly assign very low birth weight infants to receive feeds fortified according to standard, target or BUN adjustable fortification methods until the end of the feeding intervention. Feedings will be prepared in milk preparation rooms to ensure caregivers and outcomes assessor remain blinded to feeding allocation. Growth, morbidities, and nutrient intakes will be determined throughout hospitalization and skinfolds assessed at 36 weeks. At 4 months CA, growth and body composition will be determined by air displacement plethysmography on a subset of infants. Neurodevelopment will be assessed using the Bayley Scales of Infant and Toddler Development, at 18-24 months CA.

DETAILED DESCRIPTION:
The end of the feeding intervention is defined as: the infant is 36+0 weeks CA, is discharged home, or receives two oral feeds daily for three consecutive days without top-up. The exception to the 36+0 weeks intervention end-date is in the situation where an infant remains hospitalized but has not completed at least four weeks of the feeding intervention (i.e. 4 weeks following Study Day 1).

ELIGIBILITY:
Inclusion Criteria:

* ≤1250 g birth weight or Gestational Age <30+0 weeks and <1500 g birth weight.
* Parental/guardian consent to participate.
* Consent for the use of pasteurized donor milk if mother's milk is not available.

Exclusion Criteria:

* Infant received fortifier or formula before Study Day 1.
* Study Day 1 anticipated to occur after postnatal day 21.
* Infants with congenital or chromosomal anomalies or brain injury that may affect growth or neurodevelopment.
* Enrollment in any other clinical study affecting nutritional management during the feeding intervention.
* Reasonable potential that the infant will be transferred to a NICU where the study protocol will not be continued before they have completed at least 4 weeks of the feeding intervention.

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 615 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Composite Score | 18-24 months corrected age
  Bayley Scales of Infant and Toddler Development

SECONDARY OUTCOMES:
Language Composite Score | 18-24 months CA
  Bayley Scales of Infant and Toddler Development
Motor Composite Score | 18-24 months CA
  Bayley Scales of Infant and Toddler Development
Weight Gain during the intervention | Study Day 1 to 36 weeks corrected age or hospital discharge, whichever occurs first
  Change in z-score
Length gain during the intervention | Study Day 1 to 36 weeks corrected age or hospital discharge, whichever occurs first
  Change in z-score
Head circumference gain during the intervention | Study Day 1 to 36 weeks corrected age or hospital discharge, whichever occurs first
  Change in z-score
Body composition at the end of the intervention | 36 weeks corrected age
  Skinfolds
Serious Morbidity | Study Day 1 to 36 weeks corrected age or hospital discharge, whichever occurs first
  Composite of death, NEC, late onset sepsis, chronic lung disease or severe retinopathy of prematurity (ROP)
Health Economics | Study Day 1 to 36 weeks corrected age or hospital discharge, whichever occurs first
  Total cost incurred for in-hospital care
Weight at follow-up | 4 months corrected age
  z score
Length at follow-up | 4 months corrected age
  z score
Head Circumference at follow-up | 4 months corrected age
  z score
Body composition at follow-up (approximated) | 4 months corrected age
  Skinfolds
Body composition at follow-up (direct measurement) | 4 months corrected age
  Air displacement plethysmography

OTHER OUTCOMES:
Milk Type Received | Study Day 1 to 36 weeks corrected age or hospital discharge, whichever occurs first
  Type of milk consumed (i.e. parent, donor)
Energy and Nutrient Intakes of Infants | Study Day 1 to 36 weeks corrected age or hospital discharge, whichever occurs first
  Energy in kilocalories and nutrient intakes (i.e. macronutrients and micronutrients)
Maternal Diet During Lactation | Study Day 35±3
  Data on maternal diet during the first month of the intervention using the Canadian Diet History Questionnaire II

CONTACTS AND LOCATIONS:
Overall Officials: Deborah O'Connor, PhD RD, Principal Investigator — The Hospital for Sick Children; Sharon Unger, MD, Principal Investigator — Sinai Health System
Locations (20):
- Canada (20):
  - University of Alberta, Edmonton, Alberta
  - William Osler Health System-Brampton Civic Hospital, Brampton, Ontario
  - William Osler Health System-Etobicoke General Hospital, Etobicoke, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Trillium Health Partners-Missisauga Hospital, Mississauga, Ontario
  - Trillium Health Partners-Credit Valley Hospital, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - North York General Hospital, North York, Ontario
  - Humber River Hospital, North York, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - Mackenzie Health, Richmond Hill, Ontario
  - Scarborough Health Network-Centenary Hospital, Scarborough Village, Ontario
  - Scarborough Health Network-General Hospital, Scarborough Village, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health Toronto-St Michaels Hospital, Toronto, Ontario
  - Sinai Health System-Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - University of Toronto, Toronto, Ontario
  - Unity Health Toronto-St Josephs Health Centre, Toronto, Ontario

REFERENCES:
- [Derived] Beggs MR, Pichardo D, Chrzaniecki A, Kotsopoulos K, Bishara R, Ng E, Tomlinson C, Campbell D, Vaz S, Kiss A, Unger S, O'Connor DL. MaxiMoM InForM: individualised fortification of human milk for very low birthweight infants- protocol of a three-arm randomised clinical trial. BMJ Open. 2025 Oct 5;15(10):e105609. doi: 10.1136/bmjopen-2025-105609. PMID 41047263